

nt Registrar (Academic)

# UNIVERSITY OF THE PUNJAB

Quaid-i-Azam Campus, Lahore - Pakistan

Tele : Off. 92-42-9231106 Fax : Off. 92-42-9231103

No. D/ 8570 /Acad., Dated: 20-11- /2020.

Ms. Quratulain, Ph.D. Scholar, Institute of Social & Cultural Studies, University of the Punjab, Lahore.

The Advanced Studies & Research Board at its meeting held on 14-10-2020 approved the synopsis of your thesis titled "Effectiveness of Thinking Healthy Program for prevention of antenatal depression to improve maternal health, Pakistan" for Ph.D. research in the subject of Public Health. Dr. Javeria Saleem, Assistant Professor, Institute of Social & Cultural Studies, University of the Punjab, Lahore has been appointed as your Research Supervisor. Further, you will submit your Ph.D. thesis upto 19-10-2020. The approval of synopsis of Ph.D. scholar is subject to the grant of extension by the Advanced Studies & Research Board.

During the course of your studies, you will be desired to comply with the rules of Doctoral Programme, which are available from the office of the undersigned/DPCC.

Assistant Registrar (Academic) for Registrar



# Institute of Social & Cultural Studies



## University of the Punjab

Quaid-i-Azam Campus Lahore (54590) Pakistan Phone: 92-42-99233126, Fax: 92-42-35952998

233126, Fax: 92-42-35952998

233126, Fax: 92-42-35952998

Sulful of Social & Cultural Stude

Sulful of Social & Cultural Stude

Sulful of Social & Cultural Stude

Linkversity of the Punish

This is to inform you that Ms. Qurat UI Ain, Roll No. 14 (2014-19) has presented her synopsis in the meeting of Departmental Doctoral Program Committee (DDPC) was held on 19<sup>th</sup> December, 2019.

The DDPC approved her synopsis titled: "Effectiveness of Thinking Healthy Program for the Prevention of Antenatal Depression to Improve Maternal Health" and supervisor: "Dr. Javeria Saleem" for her dissertation.

Prof. Dr. Rubeena Zakar Director

Chairperson, DPCC



#### 1.8-12 20 DEPARTMENT OF ZOOLOGY UNIVERSITY OF THE PUNJAB

Prof. Dr. Javed Iqbal Qazi

Ref.

Dated

# BIOETHICAL CLEARANCE CERTIFICATE

Name of Ph.D Scholar:

Quratulain Ahsan

Title of Thesis:

"Effectiveness of Thinking Healthy Program for prevention of antenatal depression to improve maternal health,

Pakistan"

Name of Department:

Institute of Cultural and Social Sciences

Nature of work

- Experimental work
- Acquisition and analysis of data
- Sampling of human tissue
- Literature

#### Remarks:

It is certified that this research does not involve any hazardous experimental work. Standard ethical considerations as they are applied in this country for animal handling, animal room facilities and post-operative care will be followed. The research has no obvious negative impact on environment, human, animal and plant life.

Prof. Dr. Javed Iqbal Qazi

Convener Den Bioethics Committee

Quaid-i-Azam Campus, Lahore-54590, Pakistan Ph: 92-42 99231246, E-mail: zoology\_department\_pu@yaho

# Effectiveness of Thinking Healthy Program for prevention of antenatal depression to improve maternal health, Pakistan

#### **Background of Study:**

Postpartum depression is a major health issue for many women from diverse cultures, yet it remains underdiagnosed and undertreated, especially in low income countries. The prevalence rate of developing countries ranges from being equal to double from that of the developed world (Cooper et al., 2009). Pakistan has the highest prevalence amongst Asian countries that is 28%- 63%. More than half of the cases in Pakistan go unrecognized (Tikmani, Soomro, Tikmani, Zulfiqar, & Bhutto, 2016). Antenatal depression may complicate up to 10–37 % of pregnancies, while as many as 27–54 % of pregnancies are complicated by antenatal anxiety. Depression in pregnancy and postpartum is associated with significant morbidity (Williams et al., 2016).

# **Statement of the problem:**

In 2015, approximately 5,500,000 babies were born in Pakistan, or around 14,900 every day. Among young women (aged 20-24), 8 percent gave birth by age 18 years. Approximately 671 babies will die each day before reaching their first month, about 665 stillbirths occur every day. In Pakistan, the main causes of neonatal deaths in 2015 were prematurity (39.3 percent) (Unicef, 2015). Mood disorders in pregnancy and post-partum period are common and considered as a public health issue. Out of the meager health budget of Pakistan, only 0.4% is allocated to mental health (World Health Organization, 2009).

Preterm birth, a primary obstacle to the World Health Organization's Sustainable Development Goal 4, which is to reduce childhood mortality. The aim of the present study is to test the intervention in targeted group of pregnant women. We will hypothesize that primary care attendees can provide intervention that would show greater reductions in symptoms of depression, post-traumatic stress, and functional impairment and reduced symptoms of depressive disorder after treatment and at 3-month follow-up compared with base scores.

# Aim & Objectives of the Study:

## Study design:



### **Study Period:**

The present study will take about six months in data collection.

#### **Inclusion criteria:**

The eligibility criterion will be women who will deliver a baby with age 18-45 years, and will in the 24<sup>th</sup> -26<sup>th</sup> months of pregnancy. Interested participants will be given detailed information about the study. Informed consent will be obtained to participate in the study.

#### **Exclusion criteria:**

Women will be diagnosed serious medical condition requiring inpatient or outpatient treatment, pregnancy-related illness (except for common conditions, such as anaemia), substantial physical or learning disability or other form of psychosis will be excluded from study. Women younger than 18 and greater than 45 years will also be excluded.

.

#### Schema:

#### SCREENING FOR ELIGIBILITY OR EXCLUSION AND BASELINE ASSESSEMENTS

#### All women who attend

#### Gynae/Obs OPD - Antenatal desk



# 5.4.1 CONSORT flow diagram:



**Primary outcome of this study** is to evaluate the impact of a novel psychosomatic antenatal programme THP, meant to decrease symptoms of depression in the fourth week after childbirth. Secondary outcome is to assess the perceived level of social support, problems for which the person seeks help and women empowerment after intervention.

.

Table: Description of intervention sessions

| Sessions | Active ingredient | Timing of session delivery | Recipients |
|---|---|---|---|
| Session 1: Psycho-<br>education and Stress<br>Management | Psycho-education (Knowledge about anxiety disorders and stress management skills) | Fortnightly | All participants recruited into the intervention and their family members |
| Session 2: Personal Wellbeing | Thought challenging and behavior activation (Strategies for improving overall wellbeing, including diet, rest, relaxation, sleep, and managing common complaints during pregnancy) | Fortnightly | All participants |
| Session 3: Social | Thought challenging and behavior activation | Fortnightly | All participants recruited into the |

| Support | (Strategies for improving interpersonal relationship and social support). | | intervention and their family members |
|---|---|---|---|
| Session 4: Bonding with the infant during pregnancy | Thought challenging and behavior activation (Strategies for improving bonding with the infant during pregnancy). Addressing fear of child-birth (knowledge and planning of safe delivery). | Fortnightly | All participants recruited into the intervention |
| Booster sessions (depending on time of enrollment) | Behavior activation and problem management skills | Booster sessions will be coordinated with the recipients' routine antenatal visits | All participants recruited into the intervention |
| Session 6: Preparing for the baby and early postnatal period | Addressing fear of child-birth (strategies for planning for baby's arrival). Psychoeducation (coping with early post pregnancy challenges) | Late pregnancy | All participants recruited into the intervention arm and their family members. |

## Statistical analysis:

Quantitative data were analyzed with SPSS 21. Statistics will be compiled for the interventional group on EPDS, social support, stress, couple relationship and postpartum variables (women's somatic symptoms, childbirth outcomes). Group differences in baseline characteristics will be examined using chi-square tests, the Mann–Whitney test or the Kolmogorov-Smirnov test. Categorical data of principal variables will be presented as percentages and comparisons made by chi-square tests. Univariate analysis used average and standard deviation by 95% confidence interval. Analysis of secondary variables paired sample student *t* test will be applied.